CLINICAL TRIAL: NCT00613925
Title: Comparison of Pain Experienced by Patients Undergoing Endometrial Biopsy by Pipelle and Explora Curette
Brief Title: Endometrial Biopsy Instrument Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, MD MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OHSU RES 4145
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Pain
Keywords: endometrial biopsy; pain management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pipelle Group (Active Comparator): Women were randomized to have an endometrial biopsy collected using Pipelle de Cornier instrument.
  Interventions: Device: Pipelle de Cornier
- Explora group (Active Comparator): Women were randomized to have an endometrial biopsy collected using Explora curette instrument.
  Interventions: Device: Explora curette

INTERVENTIONS:
Device: Pipelle de Cornier — A flexible suction cannula 23.5 cm in length with an inner diameter of 2.6 mm and an outer diameter of 3.1 mm. It has a 2.4mm diameter opening on the distal end, on one side of the cannula. It is a disposable polypropylene sheath with an inner plunger and is used for blind endometrial biopsy.
  Other Names: Pipelle
  Arms: Pipelle Group
Device: Explora curette — The curette has an outer diameter of 3.0 mm and is slightly more rigid. This cannula has a sharp Randall-type cutting edge on the distal end, on one side of the cannula.
  Other Names: Explora
  Arms: Explora group

SUMMARY:
The purpose of this study is to determine the level of pain women experience during an endometrial biopsy and the effect that the biopsy tool might have on that pain. The investigators will also evaluate the adequacy of the sample each endometrial biopsy tool collects.

DETAILED DESCRIPTION:
Is there a difference in pain perceived by patients undergoing endometrial biopsy via the Pipelle or Explora curette? Currently, the instrument selected for endometrial biopsy is solely dependent on provider preference. This study aims to elucidate advantages and/or disadvantages of the Pipelle versus the Explora curette in terms of pain perceived by the patient, adequacy of sample, and provider ease of use to better aid in the selection of the appropriate device.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 and over who present to the Oregon Health and Science University Center for Women's Health and the Portland Veteran's Affairs Medical Center with an indication for endometrial biopsy, are literate in English or Spanish, who are willing to participate in the study.

Exclusion Criteria:

* Pregnancy, known or suspected
* Known cervical stenosis
* History of Mullerian tract anomalies
* History of uterine or cervical surgery
* Pelvic inflammatory disease (current or within the past 3 months)
* Sexually transmitted diseases (current)
* Puerperal or post abortion sepsis (current or within the past 3 months)
* Purulent cervicitis (current)
* Known clotting disorder
* Known uterine anomalies or fibroids distorting the cavity in a way incompatible with office endometrial biopsy
* Allergy to any component of the Pipelle or Explora curette
* Patients who are premedicated with analgesics or misoprostol
* Patients who require mechanical cervical dilation or receive paracervical block

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Portland Veterans Affairs Medical Center, Portland, Oregon

REFERENCES:
- [Result] Leclair CM, Zia JK, Doom CM, Morgan TK, Edelman AB. Pain experienced using two different methods of endometrial biopsy: a randomized controlled trial. Obstet Gynecol. 2011 Mar;117(3):636-641. doi: 10.1097/AOG.0b013e31820ad45b. PMID 21343767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2008 to August 2009; Academic outpatient OB/GYN clinic
Pre-assignment Details: 73 women enrolled; 3 excluded (1 cervical stenosis;1 had to have another procedure; 1 biopsy not indicated)
Groups:
- Pipelle Group: Women were randomized to the Pipelle for endometrial biopsy
- Explora Group: Women were randomized to the Explora device for endometrial biopsy
Period: Overall Study
Arm/Group | Pipelle Group | Explora Group
Started | 37 | 33
Completed | 37 | 32
Not Completed | 0 | 1
Not completed — 1 did not tolerate outpatient biopsy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pipelle Group | Explora Group | Total
Number analyzed (Participants) | 37 | 33 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 33 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (7.3) | 46.1 (7.7) | 45.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 33 | 70

OUTCOME MEASURES:

1. Primary Outcome: Compare Pipelle and Explora Curette Groups With Respect to Patient Perception of Pain Associated With the Procedure as Rated by a 100mm Visual Analog Scale (VAS).
Description: The 100mm Pain Visual Analog Scale (VAS) is an instrument used to capture subjective attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of pain by indicating a position along a 100mm continues line: pain scores can range from 0="No Pain" (furthest point to the left) to 100="Worst Pain in My Life" (furthest point to the right).
Time Frame: 2 minutes after biopsy procedure
Population: To demonstrate a 20 mm difference on the 100 mm visual analog scale, sample size of 35 women in each group (80% power, 0.05 alpha, SD 30mm)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pipelle Group | Explora Group
Number analyzed (Participants) | 37 | 32
mm | 62.1 (24.1) | 69.1 (28.8)

2. Secondary Outcome: Sample Adequacy
Description: adequacy of sample obtained for examination by a pathologist
Time Frame: at time of biopsy
Measure: Number; unit: percentage of participants
Arm/Group | Pipelle Group | Explora Group
Number analyzed (Participants) | 37 | 32
percentage of participants | 91.2 | 98.6

ADVERSE EVENTS:
Arm/Group | Pipelle Group | Explora Group
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33

LIMITATIONS AND CAVEATS:
Providers not blinded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No